CLINICAL TRIAL: NCT06628414
Title: Transcranial Direct Current Stimulation (tDCS) for Tinnitus - Effects of Multiple Treatment Sessions: a Randomised-controlled Pilot Study
Brief Title: WHITBY: Working Towards Better Healthcare Interventions for Tinnitus: a Brain Stimulation studY
Acronym: WHITBY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Magdalena Sereda, Assistant Professor, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 194-0524
Record Dates: First submitted 2024-09-27; First posted 2024-10-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Tinnitus
Keywords: tinnitus; brain stimulation; neuromodulation; transcranial direct current stimulation
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Double-blind, parallel, randomised, sham-controlled pilot trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial Direct Current Stimulation (tDCS) (Experimental): TDCS will be delivered using a NeuroConn DC Stimulator Plus via two 35cm2 rubber electrodes covered in saline-soaked sponges. The anode electrode will be positioned over EEG 10-20 coordinate F4 and the cathode over F3. The current will be delivered at 2mA for 20 minutes with ramp-up and ramp-down of 10 seconds. Each participant will receive 10 daily stimulation sessions over 2 weeks.
  Interventions: Device: transcranial Direct Current Stimulation
- Sham (Placebo Comparator): Same as intervention arm but the current will be delivered at 2mA for 30 seconds, after which the stimulation will be discontinued.
  Interventions: Device: transcranial Direct Current Stimulation

INTERVENTIONS:
Device: transcranial Direct Current Stimulation — transcranial Direct Current Stimulation

SUMMARY:
Tinnitus - the awareness of sound without any outside source - affects around 15% of people and can cause anxiety and depression. Treatment options are limited and do not address tinnitus directly (e.g., reduce its loudness). To do that, we must change brain activity causing tinnitus. Low-dose electrical stimulation, using a technique called transcranial Direct Current Stimulation (tDCS), is a promising approach. The technique is safe and easy to administer. Several small studies have tested tDCS for tinnitus showing some benefits.

To assess whether these benefits will generalise to other patients, we need to conduct a randomised controlled trial - a large, rigorously controlled experiment based on prior agreed procedures. Clinical trials are expensive and time-consuming to run and thus require meticulous pilot work to establish the most effective treatment regimens and the most sensitive measures of treatment outcome. The current study aims to provide such pilot information for a clinical trial of tDCS treatment of tinnitus. Using a total of 40 patients, we will establish how to best to administer tDCS and measure resulting changes in tinnitus perception and associated brain activity.

The current study is a crucial first step towards determining whether or not tDCS can effectively treat tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Suffering from subjective idiopathic tinnitus
* Sufficient understanding of English to be able to provide informed consent
* Able to safely undergo tDCS

Exclusion Criteria:

* Aged under 18
* Not suffering from tinnitus or suffering from objective tinnitus
* Insufficient understanding of English to be able to provide informed consent
* Unable to safely undergo tDCS as assessed by tDCS Safety Questionnaire
* Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Proof of concept | Assessed at study end (anticipated as 1 year after study start)
  Measured by protocol compliance and attrition

SECONDARY OUTCOMES:
Tinnitus symptom severity | Before first intervention session, after final intervention session and at 3-month follow-up
  Measured by Tinnitus Functional Index (TFI); maximum score: 100, higher score indicates greater tinnitus symptom severity
Tinnitus loudness | Before first intervention session, after each intervention session and at 3-month follow-up (VAS). Before first intervention session and after final intervention session (loudness matching)
  Measured by 10-point visual analogue scale, higher score indicates higher tinnitus loudness and by audiometric tinnitus loudness matching, with higher dB indicating higher loudness
Depression | Before first intervention session, after final intervention session and at 3-month follow-up
  Measured by Patient Health Questionnaire (PHQ-9) scores can range from 0 to 27 with a higher score indicating more severe symptoms
Anxiety | Before first intervention session, after final intervention session and at 3-month follow-up
  Measured by Generalised Anxiety Disorder Assessment (GAD-7) scored from 0 to 21, with a higher score indicating more severe anxiety
Treatment satisfaction | After final intervention session and at 3-month follow-up
  Measured by Short Assessment of Patient Satisfaction (SAPS) scores can range from 0 to 28 with higher scores indicating greater satisfaction
Adverse effects | After each intervention session (10 sessions over 2 weeks)
  Measured by in-house adverse effects questionnaire without numerical scoring system.
Electrophysiological brain activity | Before first intervention session and after final intervention session (1st and 10th of 10 sessions over 2 weeks)..
  Spontaneous oscillatory and auditory-evoked brain activity and coherence will be measured using 32-channel EEG. We will acquire basic structural brain images on a subset of 10 representative subjects to test the feasibility of creating individualised head models for EEG source imaging and tDCS current flow modelling.

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Sereda, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No